CLINICAL TRIAL: NCT03493555
Title: Optimizing PrEP Adherence for YMSM Through the Exploration of Facilitators and Barriers and by the Provision of a Culturally-Tailored Peer Navigation Program
Brief Title: Optimizing PrEP Adherence for Young Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Douglas Krakower, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 938125
Record Dates: First submitted 2018-02-08; First posted 2018-04-10 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Pre-Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Development (Experimental): Peer Health Navigator for PrEP
  Interventions: Behavioral: Peer Health Navigator for PrEP

INTERVENTIONS:
Behavioral: Peer Health Navigator for PrEP — Peer health systems navigator to improve adherence to PrEP

SUMMARY:
The specific aims of this study are:

1. To explore perceived facilitators and barriers to initiating and adhering to HIV PRE-EXPOSURE PROPHYLAXIS (PrEP) among at-risk YOUNG MEN WHO HAVE SEX WITH MEN (YMSM).
2. To assess the acceptability and feasibility of a culturally-tailored peer navigator program to optimize adherence to PrEP among YMSM.

DETAILED DESCRIPTION:
New HIV infections occur at a disproportionately high rate among young men who have sex with men (YMSM).Oral pre-exposure prophylaxis (PrEP) can reduce HIV acquisition among MSM over 90% when adherence levels are high, and increasing the effective use of PrEP among YMSM is one of the highest priorities in HIV prevention. However, YMSM face multiple barriers to initiating and adhering to PrEP, including structural barriers (e.g. housing insecurity), psychosocial factors (e.g. substance use, depression), underestimation of their risk for acquiring HIV, and ambivalence about using PrEP due to medical mistrust. In an open-label study of PrEP use by 200 YMSM, only one-third of participants had protective levels of drug in their blood at 1 year despite intensive adherence counseling, and HIV incidence was high at 3% per year. When PrEP is prescribed to YMSM in care settings, where adherence support is less intensive than in clinical studies, adherence levels, and thus effectiveness, are likely to be even lower. Without strategies to optimize adherence to PrEP for these youth, PrEP is unlikely to have a major impact on HIV incidence for YMSM.

One approach to overcoming the multi-factorial barriers that prevent YMSM from adhering to PrEP is the use of peer health system navigators. Navigators are healthcare workers who are trained to support adherence and retention in care for individuals who are at risk for suboptimal adherence. For YMSM who use PrEP, peer navigators could support adherence by connecting youth with resources to address their unmet structural and psychosocial needs and by helping them to negotiate the complexities of healthcare systems. An NICHD-funded study conducted in Boston (SMILE: Strategic Multisite Initiative for the Identification, Linkage and Engagement in Care of Youth with Undiagnosed HIV) found that peer navigation was highly acceptable for newly diagnosed HIV-infected youth, so it is likely that YMSM will find peer navigation to be acceptable for PrEP. As navigators have been used for over a decade to improve adherence in HIV-infected persons, and an evaluation showed that HIV-infected persons who used navigators had higher rates of virologic suppression, it is important to test whether peer navigation can optimize adherence to PrEP for YMSM.

Our long-term goal is to optimize adherence to PrEP for YMSM and thus decrease HIV incidence. The objective of this study, the first step towards our goal, is to develop and pilot test a peer navigator program to optimize adherence to PrEP for YMSM. We will recruit at-risk YMSM from an LGBTQ Youth-focused community health center with PrEP expertise, the Sidney Borum Jr. Health Center. The Borum Center provides care to 1200 YMSM aged 12-29 annually, half of whom are Black or Latino and 20% of whom are homeless. As incidence rates for HIV (2%) and syphilis (9%) in 2015 were over 20 and 100-fold higher at this center than in the general Boston population, and its clinicians initiate PrEP for 3-4 YMSM monthly, the Borum Center is an ideal setting to explore adherence to PrEP among the highest risk YMSM. Our specific aims are:

Aim 1. To explore perceived facilitators and barriers to initiating and adhering to PrEP among at-risk YMSM. We will conduct in-depth qualitative interviews with 32 YMSM at the Borum Center, including 8 youth who have not yet discussed PrEP with clinicians, 8 who have declined PrEP when offered by clinicians, 8 who have been adherent to PrEP, and 8 with suboptimal adherence. Discussions will include in-depth exploration of YMSM attitudes and intentions regarding PrEP and PrEP peer navigators. We will use purposive sampling to recruit a diverse sample with respect to race, ethnicity, and age, including youth who are minors.

Aim 2. To assess the acceptability and feasibility of a culturally-tailored peer navigator program to optimize adherence to PrEP among YMSM. A PrEP peer navigator program will be adapted from the SMILE study and will be informed by our findings from Aim 1. We will pilot test the program for acceptability and feasibility with 15 YMSM who are newly initiating PrEP at the Borum Center. Secondary outcomes include retention in PrEP care and adherence to PrEP, as measured by dried blood spot testing, at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15-24
* Self-identify as men who have sex with men
* Self-identify as sexually active
* Able to understand English

Exclusion Criteria:

* None

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Peer Navigation for PrEP Acceptability and Feasibility | up to 6 months post-enrollment
  For the primary outcome, the investigators will conduct qualitative interviews (using an IRB-approved semi-structured interview guide) at 3 and 6 months post-enrollment. Additionally, a question about acceptability of the intervention will be asked at 3 and 6 months post-enrollment. An affirmative response rate of 70% or higher will indicate acceptability of the intervention.

SECONDARY OUTCOMES:
PrEP Adherence Through DBS | up to 6 months post-enrollment
  For the secondary outcome, the investigators will use dried blood spot testing (DBS) to measure participants' PrEP drug levels.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Krakower, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- The Fenway Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT03493555/ICF_000.pdf